CLINICAL TRIAL: NCT03713918
Title: Clinical Assessment of Retention, Patient Satisfaction and Recurrent Caries of Endocrowns Versus Post Retained Crowns Using Reinforced Lithium Silicate.
Brief Title: Clini Asses of Retentn,Pt Satisfactn and Recurrent Caries of Endocrs Versus Post Crs Using Reinforced Lithium Silicate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sireen Taher Meheshi, Assistant lecturer,fixed prosthodontic department,faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-10-18
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: Patients requiring posterior single crowns or endocrowns
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessor will be blinded to avoid performance, detection and analysis bias. Only main investigator will be aware of the allocated patients in each group and the specific type of intervention given to every patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforced lithium silicate endocrown (Experimental): Device: Endocrown restoration
  Interventions: Other: Reinforced lithium silicate endocrowns
- Reinforced lithi silicate crn e post (Active Comparator): Device: Post retained reinforced lithium silicate crowns
  Interventions: Other: Post retained reinforced lith silicate crn

INTERVENTIONS:
Other: Reinforced lithium silicate endocrowns — The endodontically treated tooth will be impressed, and an endocrown restoration will be manufactured with reinforced lithium silicate and cemented with self adhesive cement
  Other Names: endocrowns
  Arms: Reinforced lithium silicate endocrown
Other: Post retained reinforced lith silicate crn — The endodontically treated tooth will receive a fiber post cemented with self adhesive cement and after this, the tooth will be impressed and reinforced lithium silicate crown will be cemented with self adhesive cement.
  Arms: Reinforced lithi silicate crn e post

SUMMARY:
Coronal retention of the restoration of RCT teeth is usually compromised, thus intraradicular posts combined or not with core material may be required.

The drawbacks of the conventional treatment created a necessary demand to have alternative treatment options. Among these options is the endocrown restoration. The pulpal chamber cavity provides retention and stability. Its trapezoidal shape in mandibular molars and triangular shape in maxillary molars increase the restoration's stability. The saddle form of the pulpal floor increases stability. This anatomy, along with the adhesive qualities of the bonding material, make no need for additional preparation or further use of post-involving root canals.

DETAILED DESCRIPTION:
Aim of the study:

The aim of this study is to evaluate the effect of using reinforced lithium silicate endocrowns on the recurrent caries, patient satisfaction and retention in comparison to post retained reinforced lithium silicate crowns.

The study is held to evaluate recurrent caries,patient satisfaction and retention of endodontically treated teeth restored with Endocrowns versus Post Retained Crowns using Reinforced Lithium Silicate after one year follow up .

The clinical performance of ceramic endocrowns showed a survival rate of 99 % and the success rate of 89.9 % in a 10 year retrospective study done by Bellflamme et al. 2017.

Endocrowns; a recently developed line of treatment, take the advantage of the rapidly growing discipline of adhesion to glass ceramics. As the retention and recurrent caries are decisive factors in the prognosis of a restoration' they have to be thoroughly investigated.

Patients with endodontically treated lower first molars will be collected.after teeth preparation to receive endocrowns and crowns ,secondary impressions will be taken .The Patients will be divided randomly into two groups .One group will receive reinforced Lithium Silicate Endocrowns (intervention)and the other group will receive reinforced Lithium Silicate Crowns (control) retained with fiber posts.

ELIGIBILITY:
Inclusion Criteria:

* • Patient age range of 18-55 years.

  * Patients physically and psychologically able to tolerate conventional restorative procedures.
  * Co-operative patients approving to participate in this trial.
  * Patients with root canal treated lower first molars requiring full coverage restoration.
  * Patients willing to return for follow-up examinations and assessments.
  * Endodontically treated teeth with absence of clinical diagnosis of periapical pathosis, fistula, swelling of periodontal tissues, abnormal tooth mobility and history of sensitivity to pressure

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth.
* Patients with poor oral hygiene.
* Disabilities which will not be cooperative patient for the study.
* Systemic diseases or severe medically compromised patients as uncontrolled diabetes or oral cancer.
* Patients suffer from parafunctional habits
* Teeth with fractured roots
* Teeth with lesions extending apical to the cemento-enamel junction
* Poor oral hygiene.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrent caries | one year
  It will be assessed using United States public health service (USPHS) criteria.

SECONDARY OUTCOMES:
Patient satisfaction | one year
  Questionnaire regarding patient satisfaction will be evaluated by the assessor
Retention | one year
  retention of the two groups will be assessed using the modified United States public health service (USPHS) criteria (Alpha,Bravo,Charlie)

IPD SHARING:
Plan to Share IPD: No